CLINICAL TRIAL: NCT01216241
Title: A Single Center, Double-Blind, Randomized, Comparative Study to Evaluate the Efficacy and Safety of Daptomycin Versus Placebo in Patients With Neutropenia and Fever.
Brief Title: Daptomycin Versus Placebo in Patients With Neutropenia and Fever
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has shown futility and the objectives could not be reached without enrolling a very large number of subjects.
Sponsor: University of Rochester (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Robert Betts, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAPNEUT
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Daptomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daptomycin (Active Comparator): Daptomycin intravenous 8mg/kg once per day 5-10 days.
  Interventions: Drug: Daptomycin
- Saline Placebo (Placebo Comparator): Saline solution
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Drug: Daptomycin — 8 MG/KG IV
  Other Names: Cubicin
  Arms: Daptomycin
Other: Saline Placebo — 50 ml normal saline once daily
  Arms: Saline Placebo
Drug: Daptomycin — 8 mg/kg once daily
  Other Names: Cubicin
  Arms: Daptomycin

SUMMARY:
The purpose of this study is to evaluate the benefits and side effects of daptomycin compared to placebo for the treatment of neutropenic fever.

DETAILED DESCRIPTION:
To determine whether the percentage of neutropenic subjects that become afebrile by five days after fever first develops is higher when daptomycin compared to placebo is added at the same time as anti gram-negative therapy. The five day time point is selected because it is at this point where it is recommended to add antifungal therapy to the treatment regimen if the patient is still febrile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the above categories who are currently undergoing chemotherapy.
2. Patients at least 18 of age.
3. Patient expected to reach an absolute granulocyte count of <100 cells/mm3
4. Patients who have given written consent because of the above criteria must have at least one temperature of greater or equal to 38.3° or temperatures > 38o on at least two occasions before study drug is administered.

Exclusion Criteria:

1. Patients with lymphoma or with solid tumor undergoing initial chemotherapy. Their neutropenia is of insufficient duration for adequate test of the value of an anti-gram positive antibiotic.
2. Patients undergoing auto-transplantation, for the same reason as above.
3. Patients with evidence of a clinical infection such as presence of a pulmonary infiltrate by x-ray or clinical evidence for the presence of cellulitis.
4. Patients who have received daptomycin in the two weeks prior to enrollment.
5. Patients with concomitant use of vancomycin.
6. Patients with creatinine clearance < 30 ml/min or CPK > 3x normal
7. Patients with significant hepatic dysfunction, defined as baseline liver function tests > 5x above normal.
8. Patients with known allergy to daptomycin.
9. Patients previously in this study.
10. Women of child bearing age who are either lactating or pregnant (as evidenced by a positive urine pregnancy test or positive serum beta-HCG).
11. Patients previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Betts, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on 14April2011 and last subject enrolled was 01November2012. All subjects were enrolled as inpatients at University of Rochester Medical Center.
Pre-assignment Details: All subjects, once consent was obtained were considered enrolled. If they developed a fever they were then randomized to study drug or placebo. If they did not develop neutropenic fever they did not receive study drug or placebo.
Groups:
- Daptomycin: Daptomycin intravenous 8mg/kg once per day 5-10 days.
  Daptomycin : 8 mg/kg once daily
  Daptomycin : 8 MG/KG IV
- Saline Placebo: Saline solution
  Saline Placebo : 50 ml normal saline once daily
  Daptomycin : 8 mg/kg once daily
Period: Overall Study
Arm/Group | Daptomycin | Saline Placebo
Started | 18 (18 subjects randomized. All didn't receive study drug/placebo if they didn't have neutropenic fever) | 18 (18 subjects randomized. All didn't receive study drug/placebo if they didn't have neutropenic fever)
Completed | 18 (Reporter remains blinded so the 4 completed could have been either study drug or placebo.) | 18 (Reporter remains blinded so the 4 completed could have been either study drug or placebo.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Saline Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Afebrile Neutropenic Subjects
Description: To determine whether the percentage of neutropenic subjects that become afebrile by five days after fever first develops.
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Daptomycin | Saline Placebo
Number analyzed (Participants) | 4 | 6
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Daptomycin | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/18
Other Adverse Events (participants affected / at risk) | 8/18 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=18) | Saline Placebo (N=18)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
elevated liver function tests (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=18) | Saline Placebo (N=18)
BK virus (Infections and infestations) | 1 (1) | 0 (0)
CVC line infection (Infections and infestations) | 1 (1) | 0 (0)
clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Worsening throat pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intermittent disorientation (Nervous system disorders) | 1 (1) | 0 (0)
Shaking (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Nervous system disorders) | 1 (1) | 0 (0)
Occasional hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Swelling to left upper extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DVT to left basilic vein (Vascular disorders) | 1 (1) | 0 (0)
Hypernatremaia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased stool (Gastrointestinal disorders) | 2 (2) | 1 (1)
Worsening nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear fullness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Increased liver enzymes (Hepatobiliary disorders) | 1 (1) | 1 (1)
Worsening psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash on chest and neck (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bruise to right arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister to arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anal fissure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bony pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
It was felt that this study had shown futility and objectives could not be reached without enrolling a very large number of subjects in a reasonable time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No